CLINICAL TRIAL: NCT05447442
Title: Adherence to the Hospital Guideline for Evaluation and Management of Preoperative Anemia in Preanesthesia Assessment Center (SIPAC), Siriraj Hospital
Brief Title: Guideline Adherence for Preoperative Anemia Management in a PAC
Status: Recruiting | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Mingkwan Wongyingsinn, MD, Principal Investigator, Siriraj Hospital
Other Study IDs: 273/2565
Record Dates: First submitted 2022-06-18; First posted 2022-07-07 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Guideline Adherence; Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group: Patients with anemia will be checked whether they would be assessed by protocol.

SUMMARY:
Anemia in surgical patients is a common seriously problem; around 40 % of patients presenting for major surgery are anemic problem. Patients with major surgery have significantly higher rates of acute blood loss. Whereas , patients with pre-operative anemia prone to be transfused blood component in pre-operative or intraoperative and postoperative periods that associated with worse outcomes , prolonged hospital stays , increased risk of morbidity and mortality . Therefore, patients undergoing major surgery should be optimization for pre-operative anemia.

In November 2021, Siriraj Preanesthesia Assessment Center (SIPAC) has developed and implemented a preoperative anemia management guideline which is one pillar of perioperative patient blood management. The objective of this guideline is to optimize red blood cell mass before patients having operation. The investigators are realize the important of pre-operative anemia of patients who undergoing elective surgery. The investigators will aim to evaluate adherence to the preoperative anemia management guideline protocol and perioperative outcomes and use the data of this study to setting guidelines for preoperative anemia evaluation and management in SIPAC of department of anesthesiology in Siriraj hospital for improving workflow and optimization before elective surgery, supporting to a reduction in blood transfusion, hospital stay, morbidity and health care costs of public health of Thailand.

DETAILED DESCRIPTION:
From World Health Organization (WHO) criteria for diagnosing anemia is hemoglobin level lower than 12 g/dL for women and hemoglobin level lower than 13 g/dL for men. The most of anemic patients caused by Iron deficiency anemia and chronic disease.

From frank S Hong that study about of prevalence and causes of preoperative anemia in elective major surgery show that preoperative anemia affects 13.9% of patients undergoing elective surgery. The most common is iron deficiency anemia 27.4%. Other common causes of anemia including underlying malignancy 18.3 %, end stage renal disease 11.5 % and other chronic disease 7.2%.

At present, there are several study about efficiency of iron therapy in pre-operative anemia that shown an increase in hemoglobin and a decrease in red cell transfusion when treated with iron therapy in 4-6 weeks. Detection of preoperative anemia should be optimized and evaluated as soon as possible at least 14 days before elective surgery.

Musallam et al. studied the prevalence and outcomes of anemia in the dataset of the American College of surgeons' National Surgical Quality Improvement Program show that anemic patients undergoing cardiac surgery & non-cardiac surgery present a higher mortality, prolonged hospital stay and more intensive care admission compared with patient non-anemic patients.

In November 2021, Siriraj Preanesthesia Assessment Center (SIPAC) has developed and implemented a preoperative anemia management guideline which is one pillar of perioperative patient blood management. The objective of this guideline is to optimize red blood cell mass before patients having operation. The investigators are realize the important of pre-operative anemia of patients who undergoing elective surgery. The investigators will aim to evaluate adherence to the preoperative anemia management guideline protocol and perioperative outcomes and use the data of this study to setting guidelines for preoperative anemia evaluation and management in SIPAC of department of anesthesiology in Siriraj hospital for improving workflow and optimization before elective surgery, supporting to a reduction in blood transfusion, hospital stay, morbidity and health care costs of public health of Thailand.

ELIGIBILITY:
Inclusion Criteria Patients who attend a preanesthesia clinic and have anemia.

Anemia defined as

1. Patients, with chronic kidney disease (CKD) stage 3+ or hematologic disease, have a hemoglobin level less than 10 g/dL; or
2. Patients other than No. 1 and have hemoglobin level less than 13 g/dL in men or a hemoglobin level less than 12 g/dL in women.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who attend a preanesthesia clinic and have anemia.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Protocol adherence | Through study completion, an average of 1 month
  The trial monitors adherence to the protocol (yes/no).

SECONDARY OUTCOMES:
Perioperative transfusion | 1 month after surgery
  Transfusion during perioperative period

CONTACTS AND LOCATIONS:
Overall Officials: Mingkwan Wongyingsinn, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided